CLINICAL TRIAL: NCT00958516
Title: A Phase 1 Study Evaluating the Phototoxic Potential of LEO 29102 Cream (2.5 mg/g, 1.0 mg/g, 0.3 mg/g, 0.1 mg/g, 0.03 mg/g) and the Cream Vehicle, Applied on Intact Skin of Healthy Male Subjects
Brief Title: Assessment of the Phototoxic Potential of LEO 29102 Cream
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Other
Other Study IDs: LEO 29102-C02; EudraCT Number 2009-011177-32
Record Dates: First submitted 2009-08-12; First posted 2009-08-13 (Estimated); Last update posted 2025-02-24 (Actual); Status verified 2013-10

CONDITIONS: Atopic Dermatitis
Keywords: volunteers
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- LEO 29102 cream (Experimental)
  Interventions: Drug: LEO 29102 cream

INTERVENTIONS:
Drug: LEO 29102 cream — LEO 29102 cream in different doses and the cream vehicle

SUMMARY:
The purpose of this trial is to evaluate the phototoxic potential of a single application on healthy skin of LEO 29102 cream in different doses.

ELIGIBILITY:
Inclusion Criteria:

* Subjects having understood and signed an informed consent form
* Male adults between the age of 18 and 65 years (both inclusive)
* Healthy subjects without signs of skin irritation on test areas (erythema, dryness, roughness or scaling)
* Subjects willing and able to follow all the study procedures and complete the whole study
* Subjects affiliated to a social security system

Exclusion Criteria:

* Females
* Males who are not willing to use a local contraception for the entire duration of the study, and refrain from fathering a child within 3 months following the study drug
* Systemic treatments which may interfere with the inflammatory reaction (e.g., corticosteroids and other anti-inflammatory drugs) within 2 weeks prior to randomisation
* Systemic or topical treatments suspected of causing photobiological reactions (e.g., tetracycline, thiazides, fluoroquinolones) within 4 weeks prior to randomisation
* Exposure to excessive or chronic UV radiation (i.e., sunbathing, solarium, phototherapy) within 4 weeks prior to inclusion or is planned during the study period
* Dark pigmentation of the skin or skin type that may, in any way, confound interpretation of the study results (skin types V and VI on the Fitzpatrick scale)
* Scars, moles, sunburn or other blemishes in the test area which may interfere with grading
* Any systemic or cutaneous disease on the test area that may confound interpretation of the study results (e.g., atopic dermatitis, eczema, psoriasis)
* Relevant history of or concurrent photo-induced or photo-aggravated disease (abnormal response to sunlight
* Subjects with a history of serious allergy, allergic skin rash or known sensitivity to any component of the investigational products
* Subjects who have received treatment with any non-marketed drug substance (i.e., an agent which has not yet been made available for clinical use following registration) within the last four (4) weeks before randomisation
* Participation in any other current interventional clinical trial based on interview of the subject
* Previously randomised in this trial
* Subjects impossible to contact in case of emergency
* Subjects known or, in the opinion of the investigator, are unlikely to comply with the Clinical Study Protocol (e.g. alcoholism, drug dependency or psychotic state)
* Subjects who are in an exclusion period in the National Biomedical Research Register of the French Ministry of Health
* Subjects under guardianship, hospitalised in a public or private institution for a reason other than research or subject deprived of freedom

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2009-09; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Phototoxic reaction according to the investigator's assessment | 5 days

SECONDARY OUTCOMES:
Clinical scoring and other skin reactions | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Director International Clinical Development, MD, Study Director — LEO Pharma
Locations (1):
- LEO Pharma investigational site, Saint-Quentin-en-Yvelines, France

IPD SHARING:
Plan to Share IPD: No